CLINICAL TRIAL: NCT05607160
Title: ELDERLY-T: A Non-interventional, Multicentre, Prospective Observational Study on the Effectiveness and Safety of Insulin Glargine 300 U/ml in Elderly Patients ≥75 Years of Age With Type 2 Diabetes
Brief Title: A Study to Observe How Insulin Glargine 300 U/ml is Working and is Tolerated in Elderly Patients ≥75 Years of Age With Type 2 Diabetes
Acronym: ELDERLY-T
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS16989; U1111-1280-6373 (Registry Identifier: ICTRP)
Record Dates: First submitted 2022-10-31; First posted 2022-11-07 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Type 2 diabetes patients >= 75 years

SUMMARY:
Primary objective:

- Glycemic control after initiation or switch to insulin glargine 300 U/ml in everyday clinical practice

Secondary objective:

- Treatment satisfaction

DETAILED DESCRIPTION:
Study duration per participant is expected to be approximately 24 weeks

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (T2DM) with oral antidiabetic drug (OAD) ± Glucagon-like-peptide-1 receptor agonist (GLP-1-RA) ± basal insulin (other than insulin glargine 300 U/ml)
* Age ≥75 years incl. patients from outpatient and inpatient care forms
* Glycohaemoglobin (Hba1c) ≥8.0% and ≤11.0%
* Inadequate glycaemic control (HbA1c), defined by the treating physician
* Ability and willingness to perform fasting blood glucose (BG) measurements themselves or with the support of third parties
* Signed consent form

Exclusion Criteria:

* Type 1 diabetes mellitus
* Age <75 years
* Contraindications to insulin glargine 300 U/ml
* Short-acting insulin in medication
* Current participation in clinical research
* Life expectancy <1 year
* Known alcohol or drug abuse
* Mini Mental State Examination Score ≤19

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Type 2 diabetes patients 75 years or older, for whom the treating physician has decided to initiate or switch to a therapy with insulin glargin 300 U/ml as part of the routine clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Proportion of participants achieving the HbA1c target value | 6 months
  Proportion of participants achieving their individual HbA1c target value (pre-defined by the treating physician) within 6 months of initiation or switch to insulin glargine 300 U/ml

SECONDARY OUTCOMES:
Absolute change in treatment satisfaction total score, from baseline to month 6 | Baseline to month 6
  Treatment satisfaction was measured using the Diabetes Treatment Satisfaction Questionnaire status (DTSQs) score
Absolute change in Diabetes-related quality of life total score, from baseline to month 6 | Baseline to month 6
  The diabetes-related quality of life was measured using the ELDERLY questionnaire
Absolute change in Geriatric Depression Scale (GDS) total score, from baseline to month 6 | Baseline to month 6
  The GDS was measured using the GDS-4 item questionnaire
Absolute proportion of participants achieving their individual HbA1c target value (pre-defined by the treating physician) within 3 months of initiation or switch to insulin glargine 300 U/ml | 3 months
Relative proportion of participants achieving their individual HbA1c target value (pre-defined by the treating physician) within 3 months of initiation or switch to insulin glargine 300 U/ml | 3 months
Absolute proportion of participants who achieve their individual fasting blood glucose (FBG) target value (pre-defined by the treating physician) within 3 months of initiation or switch to insulin glargine 300 U/ml | 3 months
Relative proportion of participants who achieve their individual fasting blood glucose (FBG) target value (pre-defined by the treating physician) within 3 months of initiation or switch to insulin glargine 300 U/ml | 3 months
Absolute proportion of participants who achieve their individual FBG target value (pre-defined by the treating physician) within 6 months of initiation or switch to insulin glargine 300 U/ml | 6 months
Relative proportion of participants who achieve their individual FBG target value (pre-defined by the treating physician) within 6 months of initiation or switch to insulin glargine 300 U/ml | 6 months
Absolute proportion of participants who achieve their individual FBG and HbA1c target values, from baseline to month 3 and 6 | Baseline to month 3 and 6
Relative proportion of participants who achieve their individual FBG and HbA1c target values, from baseline to month 3 and 6 | Baseline to month 3 and 6
Absolute proportion of patients who achieve their individual FBG or HbA1c target value, from baseline to month 3 and 6 | Baseline to month 3 and 6
Relative proportion of patients who achieve their individual FBG or HbA1c target value, from baseline to month 3 and 6 | Baseline to month 3 and 6
Absolute change in FBG (mg/dl, mmol/l), from baseline to month 3 and 6 | Baseline to month 3 and 6
Absolute change in HbA1c (%), from baseline to month 3 and 6 | Baseline to month 3 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational site, Germany, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org